CLINICAL TRIAL: NCT02631980
Title: Hepcidin Overexpression After Hepatectomy : Does Iron Supplementation Make Sense ?
Brief Title: HepciFer Study: Hepcidin Overexpression After Hepatectomy : Does Iron Supplementation Make Sense ?
Acronym: HepciFer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Eduardo Schiffer, M.D., University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 15-079
Record Dates: First submitted 2015-12-02; First posted 2015-12-16 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Anemia; Postoperative Blood Loss
Keywords: Hepcidin
MeSH Terms: conditions — Anemia; Postoperative Hemorrhage | interventions — ferryl iron; ferric carboxymaltose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV iron (Experimental): Postoperative iv iron administration (Ferinject) upon arrival in after surgery recovery room
  Interventions: Drug: IV iron
- IV placebo (Placebo Comparator): Postoperative iv placebo administration upon arrival in after surgery recovery room
  Interventions: Drug: IV placebo

INTERVENTIONS:
Drug: IV iron — Intravenous iron 15 mg/kg (max 1000 mg) in 250 ml 0.9% saline
  Other Names: Ferinject
  Arms: IV iron
Drug: IV placebo — Intravenous 0.9% saline (250 ml)
  Other Names: Placebo
  Arms: IV placebo

SUMMARY:
Hepcifer Trial is designed to assess the value of iv iron administration immediately after liver surgery and consequences of inflammation on iron balance. Fifty patients will be randomized in two treatment groups. Patients will be assigned to receive either iv iron or placebo immediately after liver resection surgery. Biological inflammation parameters, hemoglobin, serum iron and hepcidin levels will be assessed prior to surgery and at day 1, 3, 7, 15 and 30 after surgery.

DETAILED DESCRIPTION:
The iron homeostasis is now well known. Indeed, the discovery of hepcidin, a protein synthesized by the liver, has provided a better understanding of iron metabolism and the resulting anemia disruption of this homeostasis.

Although morbidity decreased hepatic surgery remains a major surgery as by surgical difficulty by support intra- and postoperatively.

A preliminary study, the investigators found that patients had preoperative anemia (oncological context) increased postoperatively, increasing the morbidity.

Few clinical studies on hepcidin and anemia were carried out, because of the difficulty of metering (mass spectrometry) as well as its cost.

In this clinical trial, the investigators plan to assess the value of iv iron administration versus iv placebo treatment immediately after liver surgery and consequences of inflammation on iron balance. In addition, an evaluation of the well being of patients will be performed postoperatively to measure the functional and psychological impact of anemia.

This is a monocentric, randomized, double blinded and placebo controlled trial. Iron iv injection will be administered postoperatively. Hematology assessments, biological iron deficiency, inflammation and coagulation will be realized pre and postoperatively. Hepcidin is assayed by an ELISA method.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled liver surgery,
* Liver resection > 2 segments.

Exclusion Criteria:

* Age below 18yrs,
* Pregnancy,
* Emergent surgery,
* Sepsis,
* Immunosuppressive therapy,
* Renal insufficiency (GFR<30ml/min/m2),
* Hypersensitivity to iron,
* Iron overload.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Hemoglobin level | Postoperative Day 7
  Blood sample at postoperative Day 7

SECONDARY OUTCOMES:
Length of hospital stay | Through study completion, an average of 1 year
Quality of life Questionnaire at day 30 | Postoperative Day 30
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Schiffer, MD, Principal Investigator — University of Geneva
Locations (1):
- University of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No